CLINICAL TRIAL: NCT01202149
Title: Bilateral Comparison Study of Elidel® (Pimecrolimus) Cream 1% and Hylatopic™ Plus Emollient Foam™ Emollient Foam in the Treatment of Subjects With Atopic Dermatitis
Brief Title: Bilateral Comparison Study of Elidel 1% and Hylatopic Plus Emollient Foam for the Treatment of Subjects With Atopic Dermatitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Frankel, Amylynne, M.D. (Other)
Collaborators: Onset Therapeutics, Inc (Unknown)
Responsible Party: Principal Investigator - Amylynne Frankel, MD, Clinical Dermatopharmacology Fellow, Mount Sinai School of Medicine, Department of Dermatology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 09-0879
Record Dates: First submitted 2010-09-14; First posted 2010-09-15 (Estimated); Last update posted 2011-04-15 (Estimated); Status verified 2011-04

CONDITIONS: Eczema; Atopic Dermatitis
Keywords: eczema; elidel; non-medicated device; hylatopic plus; pimecrolimus; bilateral comparison study; topical therapy
MeSH Terms: conditions — Eczema; Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Elidel Right Side, Hylatopic Plus Left Side (Active Comparator): Elidel applied topically on Right Side of body twice a day and Hylatopic plus emollient foam applied topically on Left Side of body three times a day
  Interventions: Device: Elidel (pimecrolimus cream, 1%) Hylatopic Plus Emollient Foam (non-medicated device)
- Elidel Left Side Hylatopic Plus Right Side (Active Comparator): Elidel applied topically on Left Side of body twice a day and Hylatopic plus emollient foam applied topically on Right Side of body three times a day
  Interventions: Device: Elidel (pimecrolimus cream, 1%) Hylatopic Plus Emollient Foam (non-medicated device)

INTERVENTIONS:
Device: Elidel (pimecrolimus cream, 1%) Hylatopic Plus Emollient Foam (non-medicated device)

SUMMARY:
This is an investigator-blinded, bilateral comparison study in 30 subjects with atopic dermatitis. It is designed to assess and compare the efficacy of Elidel® (pimecrolimus) cream 1% and Hylatopic™ Plus Emollient Foam™ in subjects with atopic dermatitis. Subjects will apply Elidel® (pimecrolimus) cream 1% twice daily for four weeks on a chosen target eczematous area located on one side of the body and then apply Hylatopic™ Plus Emollient Foam™ three times daily on a symmetrical target eczematous area on the opposite side of the body. A randomized list will be created to determine which side the subject applies each medication.

Subjects will be consented prior to any study evaluations or procedures. After signing the consent and meeting all inclusion/exclusion criteria, qualified and enrolled subjects will apply study medication (Elidel® and Hylatopic™ Plus Emollient Foam™) to chosen affected areas for four weeks. Photography will be used to record the location of target lesions at the baseline, week two and week four/final visits. Subject's disease status will be assessed by two methods: 1) Physician's Global Assessment (PGA) and 2) Target Lesion Symptom Score (TLSS) (see sections V.B.2 and V.B.3). PGA as well as TLSS will be made at baseline (Day 0), week two (Day 14 +/- 2 days) and week 4/final visit (Day 28 +/- 2days) visits for each of the target lesions. Half scales (i.e. 0.5, 1.5) will not be used. The presence or absence of skin atrophy and telangiectasias will be noted at each study visit as well.

Additionally, subjects' self-assessments of their perception of degree of disease and itching severity control will be collected at each visit for each target lesion. This assessment will be made using a four point scale and Itch Severity Scale (visual analogue score) respectively (see section V.B.4). Lastly, subjects will take a Product Preference Survey at week 4/final visit (Day 28 +/- 2days). Parents (or guardians) will moderate Product Preference Surveys for subjects that are younger than 12 years of age.

DETAILED DESCRIPTION:
This is an investigator-blinded, bilateral comparison study in 30 subjects with atopic dermatitis. It is designed to assess and compare the efficacy of Elidel® (pimecrolimus) cream 1% and Hylatopic™ Plus Emollient Foam™ in subjects with atopic dermatitis. Subjects will apply Elidel® (pimecrolimus) cream 1% twice daily for four weeks on a chosen target eczematous area located on one side of the body and then apply Hylatopic™ Plus Emollient Foam™ three times daily on a symmetrical target eczematous area on the opposite side of the body. A randomized list will be created to determine which side the subject applies each medication.

Subjects will be consented prior to any study evaluations or procedures. After signing the consent and meeting all inclusion/exclusion criteria, qualified and enrolled subjects will apply study medication (Elidel® and Hylatopic™ Plus Emollient Foam™) to chosen affected areas for four weeks. Photography will be used to record the location of target lesions at the baseline, week two and week four/final visits. Subject's disease status will be assessed by two methods: 1) Physician's Global Assessment (PGA) and 2) Target Lesion Symptom Score (TLSS) (see sections V.B.2 and V.B.3). PGA as well as TLSS will be made at baseline (Day 0), week two (Day 14 +/- 2 days) and week 4/final visit (Day 28 +/- 2days) visits for each of the target lesions. Half scales (i.e. 0.5, 1.5) will not be used. The presence or absence of skin atrophy and telangiectasias will be noted at each study visit as well.

Additionally, subjects' self-assessments of their perception of degree of disease and itching severity control will be collected at each visit for each target lesion. This assessment will be made using a four point scale and Itch Severity Scale (visual analogue score) respectively (see section V.B.4). Lastly, subjects will take a Product Preference Survey at week 4/final visit (Day 28 +/- 2days). Parents (or guardians) will moderate Product Preference Surveys for subjects that are younger than 12 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ≥ 2 years old.
* Subjects must be in good general health as confirmed by medical history and physical examination.
* Females of child-bearing potential must have a negative urine pregnancy test at the baseline visit and agree to use adequate birth control during the study (barrier, oral, injection, intrauterine). NOTE: Post-menopausal (amenorrheic for at least one year) and surgically sterile (tubal ligation and/or hysterectomy) are considered to be of non child-bearing potential.
* Diagnosis of atopic dermatitis for at least one year with symptoms on arms, trunk, and/or legs.
* Subject must have a static Investigator's Global Assessment (IGA) of at least 2 or 3 (mild-moderate severity) for each selected target lesion
* Disease must be stable or slowly worsening for more than one week prior to the Screening Visit, as reported by the subject.
* Subjects or their guardians must be able to read, sign, and date the informed consent, and abide by study restrictions for its duration.

Exclusion Criteria:

* Females who are pregnant, attempting to conceive, or breastfeeding.
* Subjects with known hypersensitivity to either study drug.
* Subjects with AD on >30% body surface area
* Subjects with overt signs of skin atrophy, telangiectasias and/or striae in the target area.
* Subjects with a current active skin malignancy or infection.
* Subjects requiring the use of medications known to alter the course of atopic dermatitis during the study treatment.
* Subjects who have received systemic antibiotics within 2 weeks.
* Subjects using systemic corticosteroids or immunosuppressants within 28 days of the Screening Visit.
* Subjects who have received topical corticosteroids or other topical therapies (tar, calcineurin inhibitors) for atopic dermatitis within 7 days of the Screening Visit.
* Subjects using phototherapy (UVB, PUVA) within 28 days of the Screening Visit.
* Subjects who are currently participating in or, with in the previous 28 days, have participated in another study for the treatment of atopic dermatitis.
* Subjects with clinical conditions that may pose a health risk to the subject by being involved in the study or detrimentally affect regular follow-up of the subject.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-03; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Improvement and maintenance of PGA, TLSS, and subjective eczema control of Hylatopic Plus Emollient Foam versus Elidel Cream | 26 weeks

SECONDARY OUTCOMES:
Improvement and maintenance of signs of eczema
  Improvement and maintenance of signs of eczema (erythema, population/infiltration, lichenification, and scaling/dryness) with twice daily Elidel applied topically to one side of the body as compared to three times days Hylatopic Plus applied topically to the other side of the body; Assessment for any clinical signs of atrophy or telangiectasia; Improvement in patient self-assessments

CONTACTS AND LOCATIONS:
Locations (1):
- Mount Sinai Faculty Practice Associates, New York, New York, United States